CLINICAL TRIAL: NCT02352285
Title: Assessment of Clinical Outcome and Treatment Quality Under Adequate Use of Tolvaptan In Correction of Hyponatremia in Patients Hospitalized With Worsening Heart Failure and Hyponatremia
Brief Title: Outcome and Treatment Quality Study of Tolvaptan to Treat Hyponatremia in Patients With Heart Failure
Acronym: AQUATIC
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Korea Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 156-KOB-1201i; NCT01865214 (obsolete NCT alias)
Record Dates: First submitted 2012-12-20; First posted 2015-02-02 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2016-11

CONDITIONS: Heart Failure With Hyponatremia
MeSH Terms: interventions — Tolvaptan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tolvaptan (Experimental): Tovaptan tablet 15mg, 30mg, 60mg, once a day, oral
  Interventions: Drug: Tolvaptan
- placebo (Placebo Comparator): placebo tablet 15mg, 30mg, 60mg, once a day, oral
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tolvaptan — Start with 15mg to titrate upwards to 30mg to 60mg, once a daily
  Other Names: Samsca
  Arms: Tolvaptan
Drug: Placebo — Start with 15mg to titrate upwards to 30mg to 60mg, once a daily
  Arms: placebo

SUMMARY:
The objective is to evaluate the efficacy and safety on the tolvaptan for increasing serum Na levels in patients with worsening heart failure and hyponatremia.

DETAILED DESCRIPTION:
This is a phase 4, multicenter, randomized, double-blind, placebo-controlled, parallel-group interventional study comparing tolvaptan (15 to 60 mg) to placebo in adult patients hospitalized (or admission to emergency room) due to worsening of heart failure and dilutional hyponatremia. All patients will be on standard therapy for heart failure.

ELIGIBILITY:
Inclusion Criteria:

1. Patients hospitalized due to heart failure with clinically significant hyponatremia (except hypovolemic) (defined as serum Na < 125 mEq/L or less marked hyponatremia that is symptomatic and has resisted correction with fluid restriction) prior to randomization.
2. Male and female patients aged ≥ 20 years.
3. New York Heart Association (NYHA) class III/Ⅳ
4. Signs of extracellular volume expansion, defined as two or more of the following: JVD, peripheral edema, dyspnea or pulmonary congestion.
5. B-type natriuretic peptide (BNP) ≥ 150 pg/mL or N terminal (NT)-proBNP ≥ 450 pg/mL.

Exclusion Criteria:

1. Women who are pregnant, breast feeding, or of childbearing potential who are not using acceptable contraceptive methods
2. Patients with hyponatremia in hypovolemic states, defined as the presence of clinical and historical evidence of extracellular fluid volume depletion
3. Patients unable to sense or respond to thirst.
4. Patients who are likely to require prolonged hospitalization for reasons other than chronic heart failure (CHF)
5. Patients with recent prior treatment for hyponatremia
6. Patients with severe hyponatremia symptoms requiring immediate intervention with hypertonic saline
7. Patients with causes of neurological symptoms, which are attributable to psychological (psychoses), structural (dementia of the Alzheimer's type, post-infarct dementia) or other metabolic causes
8. Patients with acute and transient hyponatremia associated with head trauma or severe neurological injury
9. Patients with a history of hyponatremia known to be due to severe, untreated hypothyroidism/adrenal insufficiency.
10. Patients with psychogenic polydipsia.
11. Patients with systolic BP < 90 mmHg at screening.
12. Patients with a history of hypersensitivity and/or idiosyncratic reaction to benzazepine or benzazepine derivatives (such as benazepril), or tolvaptan.
13. Patients with a history of drug or medication abuse within the 3 months prior to screening, or current alcohol abuse.
14. Patients with uncontrolled diabetes mellitus
15. Patients with a current urinary tract obstruction
16. Anuric patients.
17. Patients with a serum creatinine > 3.5 mg/dL at screening.
18. Terminally ill patients or patients with a moribund condition who have little chance of short-term survival.
19. Patients whose hyponatremia is the result of any medication that cannot safely be withdrawn, such as anti-convulsants and anti psychotics
20. Patients receiving desmopressin within 2 days of screening.
21. Patients who have participated in another investigational drug trial within the past 30 days.
22. Any patient who, in the opinion of the investigator, would not be able to comply with the study drug administration or study procedures, or whose overall medical condition would prohibit their participation in the study.
23. Patients treated and/or to be treated with strong cytochrome P450 (CYP) 3A inhibitors
24. Patients with rare hereditary problems of galactose intolerance, Lapp lactase deficiency or glucose- galactose malabsorption.
25. Patients with a AST or ALT > ULN 2.5 or total bilirubin > 2mg/dL

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Average daily AUC of change from baseline in serum Na level to day 4 within the double-blind treatment period | from baseline to day 4

SECONDARY OUTCOMES:
Average amount of furosemide used during hospitalization. | from day 1 to discharge date (up to subject condition day 2 ~ day 30)
Average amount of furosemide used during out-patient period. | from baseline to day 30 and day 60

CONTACTS AND LOCATIONS:
Overall Officials: Dongju Choi, MD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seoul, South Korea